CLINICAL TRIAL: NCT05452603
Title: Usefulness of Wireless pH Monitoring in the Diagnosis of Gastroesophageal Reflux Disease
Brief Title: Usefulness of Wireless pH Monitoring in GERD Diagnosis
Status: Completed | Type: Observational
Sponsor: Hospital de Clinicas José de San Martín (Other)
Responsible Party: Principal Investigator, Maria Marta Piskorz, Principal investigator, Hospital de Clinicas José de San Martín
Other Study IDs: 27251302710
Record Dates: First submitted 2022-07-04; First posted 2022-07-11 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Gastroesophageal Reflux
Keywords: gastroesophageal reflux disease; gray area; wireless pH monitoring
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Study group: Thirty consecutive patients with GERD symptoms and an acid exposure time (AET) measured by impedance measurement/pH between 4 and 6% will be included.
  Interventions: Device: 96-hour off IBP wireless pH monitoring capsule

INTERVENTIONS:
Device: 96-hour off IBP wireless pH monitoring capsule — The endoscopic pH measurement capsule will be placed 6cm above the squamocolumnar junction, determined endoscopically, in the sedated patient. Then the plot will be read.

SUMMARY:
Gastroesophageal reflux disease (GERD) is extremely common in our environment. Its diagnosis is complex. The Lyon Consensus defined, based on 24-hour pH monitoring, that an acid exposure time greater than 6% is definitely abnormal, less than 4% is normal, and between 4 and 6% is a gray area.

The objective of this study is to describe the change in therapeutic behavior based on the result of prolonged pH recording performed with a 96-hour wireless pH measurement capsule in patients with GERD symptoms and an acid exposure time measured by impedanciometry/pH of 24 hours in the gray area. Also, describe the therapeutic outcomes.

DETAILED DESCRIPTION:
Thirty consecutive patients with GERD symptoms and an acid exposure time (AET) measured by impedance measurement/pH between 4 and 6% will be included.

A 96-hour off IBP wireless pH monitoring capsule will be performed. The worst day, the average of the 4 days and the presence of 2 or more days with AET>6% and the 4 days with AET<4% will be recorded.

Patients will be categorized into GERD, reflux hypersensitivity, and functional heartburn. A treatment will be established based on these categories and the GERDq will be measured at 8 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age, with symptoms of gastroesophageal reflux, who have undergone a 24-hour impedance pH study without proton pump inhibitors (PPIs), whose AET is between 4 and 6% will be included consecutively. .

Exclusion Criteria:

* Patients with severe comorbidities: Liver cirrhosis, oncological disease, autoimmune diseases, cognitive impairment, psychiatric diseases, bleeding diathesis or anticoagulation
* Pregnant women
* Patients with severe esophagitis, esophageal varices, esophageal strictures, Barrett's esophagus, anti-reflux surgery
* Patients with history of pacemaker or defibrillator, since they can interfere with the signal.
* Patients with nickel allergy
* Patients that refuses to sign the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ≥ 18 years of age, with symptoms of Gastroesophageal Reflux, who have undergone a 24-hour impedance pH study without Proton Pump Inhibitors (PPIs), whose AET is between 4 and 6% will be included consecutively. .
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-06-20 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-07-20 (Actual)

PRIMARY OUTCOMES:
GERD Proportion | june 2021-june 2023
  estimate the proportion of GERD measured by wireless pH monitoring capsule in patients in the gray area
Therapeutic response | june 2021-june 2023
  To compare the GERDq scale before and after treatment with proton pump inhibitors.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Clinicas Jose de San Martin. Buenos Aires University, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided